CLINICAL TRIAL: NCT00948753
Title: Safety and Efficacy of Maraviroc, a CCR5-inhibitor in Prophylaxis of Graft-Versus-Host Disease in Patients Undergoing Non-Myeloablative Allogeneic Stem-Cell Transplantation
Brief Title: Maraviroc in Patients Undergoing Non-Myeloablative Allogeneic Stem-Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04708
Record Dates: First submitted 2009-07-23; First posted 2009-07-29 (Estimated); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Graft-versus-host Disease; Hematopoietic Stem Cell Transplantation
Keywords: Graft-versus-host disease; GVHD; Maraviroc; non-myeloablative allogeneic stem-cell transplantation; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Maraviroc; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1: 150mg Maraviroc (Experimental): 150mg twice daily
  Interventions: Drug: Maraviroc 150 MG
- Phase 1: 300mg Maraviroc (Experimental): 300mg twice daily
  Interventions: Drug: Maraviroc 300 mg
- Phase 2: 300mg Maraviroc (Experimental): 300mg twice daily
  Interventions: Drug: Maraviroc 300 mg Phase II

INTERVENTIONS:
Drug: Maraviroc 150 MG — Maraviroc b.i.d. (in addition to the standard prophylaxis therapy of tacrolimus and methotrexate) beginning after last dose of chemotherapy conditioning regimen until day 30 after stem-cell infusion.
  Other Names: CCR5 Blockade
  Arms: Phase 1: 150mg Maraviroc
Drug: Maraviroc 300 mg — Maraviroc b.i.d. (in addition to the standard prophylaxis therapy of tacrolimus and methotrexate) beginning after last dose of chemotherapy conditioning regimen until day 30 after stem-cell infusion.
  Other Names: CCR5 Blockade
  Arms: Phase 1: 300mg Maraviroc
Drug: Maraviroc 300 mg Phase II — Maraviroc b.i.d. (in addition to the standard prophylaxis therapy of tacrolimus and methotrexate) beginning after last dose of chemotherapy conditioning regimen until day 30 after stem-cell infusion.
  Other Names: CCR5 Blockade
  Arms: Phase 2: 300mg Maraviroc

SUMMARY:
This study investigates the effectiveness and safety of Maraviroc (an oral medication given twice daily given in addition to the standard GVHD prophylaxis) in preventing Graft versus Host Disease (GVHD) in patients undergoing non-myeloablative allogeneic stem-cell transplantation (SCT). Subjects will receive Maraviroc bid (in addition to standard GVHD prophylaxis) beginning after the last dose of the chemotherapy conditioning regimen until day 30 after stem-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo non-myeloablative allogeneic stem-cell transplantation.
* meet institutional eligibility criteria for allogeneic SCT. Significant criteria are:

  * Renal function: Serum creatinine <2; or calculated creatinine clearance > 40 mL/min/1.72m2;
  * Hepatic function: Baseline direct bilirubin, ALT or AST lower than three times the upper limit of normal;
  * Pulmonary disease: FVC or FEV1 > 40% predicted; Cardiac ejection fraction > 40%.

Exclusion Criteria:

* Patients not expected to be available for follow-up in our institution for at least 100 days after the transplant
* Patients who are not undergoing standard non-myeloablative SCT with Flu/Bu conditioning and Tax/MTX GVHD prophylaxis
* Patients with uncontrolled bacterial, viral or fungal infections
* Patients who take strong inducers or inhibitors of the CYP450A4
* Patients receiving other investigational drugs for GVHD
* Women who are pregnant, plan to become pregnant or are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Porter, MD, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Derived] Reshef R, Luger SM, Hexner EO, Loren AW, Frey NV, Nasta SD, Goldstein SC, Stadtmauer EA, Smith J, Bailey S, Mick R, Heitjan DF, Emerson SG, Hoxie JA, Vonderheide RH, Porter DL. Blockade of lymphocyte chemotaxis in visceral graft-versus-host disease. N Engl J Med. 2012 Jul 12;367(2):135-45. doi: 10.1056/NEJMoa1201248. PMID 22784116

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2: 300mg Maraviroc: 300mg twice daily
  Maraviroc 300 mg: Maraviroc b.i.d. (in addition to the standard prophylaxis therapy of tacrolimus and methotrexate) beginning after last dose of chemotherapy conditioning regimen until day 30 after stem-cell infusion.
Period: Phase 1
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc
Started | 7 | 6 | 0
Completed | 7 | 6 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc
Started | 0 | 0 | 25
Completed | 0 | 0 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants totaled 13 for phase I and 25 for phase 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc | Total
Number analyzed (Participants) | 7 | 6 | 25 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 15 | 26
  >=65 years | 0 | 2 | 10 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 10 | 15
  Male | 5 | 3 | 15 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 7 | 6 | 23 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 25 | 38

OUTCOME MEASURES:

1. Primary Outcome: Safety of Maraviroc
Description: number of Adverse Events following exposure to Maraviroc
Time Frame: 1 year
Population: patients receiving SCT
Measure: Number; unit: Number of AEs
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc
Number analyzed (Participants) | 7 | 6 | 25
Number of AEs | 8 | 6 | 18

2. Primary Outcome: Efficacy of Maraviroc
Description: Efficacy is measured by number of participants progressing to acute GVHD. If acute GVHD is noted in a participant following exposure to study drug, then efficacy was not achieved.
  If no GVHD was noted following exposure, then efficacy was achieved in that participant
Time Frame: 8 weeks
Measure: Number; unit: Participants
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc
Number analyzed (Participants) | 7 | 6 | 25
Participants | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetic Profile of Maraviroc in Patients Undergoing Nonmyeloablative Allogeneic SCT
Description: Plasma maraviroc levels were measured in the blood with a target level of 100 ng per milliliter. Blood was drawn on Day 0 and Day 10-12 at pre-dose, 1, 2, 3, 4, 6, and 12 hours post-dose. Data was analyzed looking at the number of patients to achieve the target of 100 ng per milliliter at any time point.
Time Frame: pre-dose, 1,2,3,4,6,12 hours post-dose
Population: not enough data was collected to reach statistical power for plasma maraviroc levels in the Phase 2 group.
Measure: Number; unit: number of patients to reach target
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc
Number analyzed (Participants) | 7 | 6 | 25
number of patients to reach target | 4 | 6 | 0

4. Secondary Outcome: Number of Patients Treated With Maraviroc During SCT That Develop Chronic GVHD
Description: count of how many patients treated with Maraviroc during SCT go on to develop chronic GVHD in 1 year
Time Frame: 1 year
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc
Number analyzed (Participants) | 7 | 6 | 25
Participants | 1 | 3 | 2

5. Secondary Outcome: Rate of Early Mortality After Transplant
Description: Number of participants who died without relapse within 1 year of SCT
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc
Number analyzed (Participants) | 7 | 6 | 25
Participants | 2 | 0 | 4

6. Secondary Outcome: Number of Participants Who Relapsed During Study Period
Description: Number of participants who received Maraviroc during SCT who relapsed within 1 year and 11 months. This was based on a diagnosis made by their physician that their primary cancer had returned.
Time Frame: 1 year and 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc
Number analyzed (Participants) | 7 | 6 | 25
Participants | 2 | 2 | 15

ADVERSE EVENTS:
Arm/Group | Phase 1: 150mg Maraviroc | Phase 1: 300mg Maraviroc | Phase 2: 300mg Maraviroc
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/25
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 17/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: 150mg Maraviroc (N=7) | Phase 1: 300mg Maraviroc (N=6) | Phase 2: 300mg Maraviroc (N=25)
Mucositis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 5 (5)
Bacteremia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (3)
Abnormal LFTs (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gout (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Septic arthritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No